CLINICAL TRIAL: NCT04384848
Title: Evaluating Patient-Reported Outcomes Monitoring in Routine Care of Patients With Chronic Myeloid Leukemia for Increasing Adherence and Clinical Response to THerapY: The EMPATHY Pilot Study
Brief Title: The EMPATHY Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Fondazione GIMEMA (Other); Augusta University (Other)
Responsible Party: Principal Investigator, David Cella, Professor, Medical Social Sciences; Feinberg School of Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R21CA230367-01A1 (NIH)
Record Dates: First submitted 2020-04-17; First posted 2020-05-12 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Leukemia, Chronic Myeloid; Cancer
Keywords: Cancer; Leukemia, Chronic Myeloid; Health-Related Quality Of Life; Patient Reported Outcome
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic myeloid leukemia (CML) patients (Experimental): CML patients undergoing first-line tyrosine kinase inhibitor (TKI) therapy
  Interventions: Other: EMPATHY Pilot

INTERVENTIONS:
Other: EMPATHY Pilot — The goal of this pilot is to develop and pilot a tailored monitoring intervention targeting symptomatic, Patient-reported adverse events (AEs) in chronic myeloid leukemia (CML) Patients undergoing first-line tyrosine kinase inhibitor (TKI) therapy. The tailored monitoring intervention will draw primarily from the PRO-CTCAE Item Library, with additional items drawn from the FACIT and EORTC Item libraries as necessary. After identifying the full set of AEs to be monitored, we will load the Patient assessment and report program into tablets for electronic administration in the busy clinic setting. We will then pilot a six-month intervention aimed to monitor and manage emerging AEs, coupled with assessment of intervention feasibility, Patient acceptability and satisfaction, provider acceptability and clinical management utility, adherence to TKI therapy, and HRQoL. We expect that adherence to therapy, clinical response, and HRQoL will be enhanced by such an intervention.

SUMMARY:
The proposed study, may significantly contribute to improve healthcare delivery in patients with Chronic Myeloid Leukemia (CML) treated with modern tyrosine kinase inhibitors (TKIs) in two ways. First, it may provide novel empirical data on the positive effects of systematically monitoring of patient-reported adverse events (AEs) in routine practice for improving symptom management and adherence to therapy. Second, it will inform the development of a large international randomized controlled trial (RCT) to test whether systematic collection of patient-reported AEs, could improve clinical response to TKI therapy.

DETAILED DESCRIPTION:
The evolution in the understanding of the biology of Chronic Myeloid Leukemia (CML), that eventually translated into highly effective molecular targeted therapies, is unparalleled in cancer medicine. This knowledge led the development of a number of orally active molecule tyrosine kinase inhibitors (TKIs) that have dramatically improved clinical outcomes. In less than two decades, the 10-year survival probability increased from 20 to 53% with previous (IFN)-therapies to about 90% in the TKI era. Life expectancy of these patients now approaches that of the general population. While oral TKIs are now the standard of care for CML, it should be considered that therapy is lifelong and patients are requested to take medication on a daily basis. Importantly, there is convincing evidence that full adherence to therapy is a critical factor to obtain and maintain an optimal response to therapy. However, non-adherence is a major challenge in CML, since side effects induced by these drugs negatively impact on patient's quality of life (QoL), seriously undermine full adherence with treatment schedule and thereby often lead to sub-optimal clinical responses to drugs. From previous Preliminary Data we extrapolated the following evidences: Systematic monitoring of Patient-Reported Outcomes (PRO) in routine care has several advantages, such as improved symptom control, enhanced patient-physician communication, as well as patient satisfaction and wellbeing. Furthermore, it was found that Adverse Events (AEs) are the most frequent cause for non-adherence to CML therapy and that even experienced physicians tend to underestimate burden of TKIs of their patients. This mismatch might have major clinical implications in disease management, as physicians might not be able to early identify those patients who might be at heightened risk of poor adherence behavior. Given these findings, we hypothesized that systematic electronic monitoring of Patient-Reported AEs in CML routine practice may improve adherence to therapy, quality of life, and clinical response to therapy. This hypothesis will be addressed in the experiments of the following Specific Aims: 1) To develop an online platform for systematic monitoring of patient-reported AE assessment that is tailored to the unique demands of TKI therapy for CML. 2) To assess patient and physician acceptability and satisfaction with use of this platform in CML routine practice and evaluate its value in improving symptom management, quality of life, adherence to therapy as well as preliminary efficacy. We anticipate this study will provide unprecedented information on the value of systematically collecting patient-reported AEs information in CML routine care. If positive, our results will inform the development of large international randomized controlled trial (RCT) to investigate whether this experimental approach can improve depth and rates of clinical responses to TKI therapies in CML patients.

Dr. Fabio Efficace is also a Principal Investigator on this study. He is also a Professor in the Department of Medical Social Sciences at Northwestern University, Feinberg School of Medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Philadelphia chromosome positive and/or BCR-ABL positive CML confirmed by cytogenetic and/or molecular analysis;
2. Newly diagnosed chronic phase (CP)-CML Patients planned to receive one of the following TKI approved as first line treatment: imatinib, dasatinib, nilotinib or bosutinib;
3. Adult Patients (≥18 years) at the time of study entry; Children under the age of 18 will be excluded from the study. The exclusion of children is justified by the following circumstances: a) The condition is relatively rare in children, as compared to adults; b) Issues of study preclude direct applicability of hypotheses and/or interventions to both adults and children.
4. Written informed consent.
5. Written informed consent from Patient's physician as a participant.
6. Newly diagnosed Chronic Phase (CP)-CML Patients who are within 4 weeks of first line TKI therapy (anyone of the TKI approved in the USA and Europe, that is: imatinib, dasatinib, nilotinib or bosutinib).
7. Ability to read/converse in English (Northwestern University and Augusta University Sites). Ability to read/converse in Italian (GIMEMA Centers).

Patient exclusion criteria will include:

1. Major cognitive deficits or psychiatric problems hampering a self-reported evaluation;
2. Having received any CML treatment - other than TKI - for more than 3 months prior to receiving current TKI therapy.

This project will focus on CML, which affect both men and women. Therefore, there are no exclusion/inclusion criteria based on sex/gender. In addition, there are no exclusion/inclusion criteria based on race and ethnicity.

Physician inclusion criteria will include:

1)Provider of clinical care for Patient who meets inclusion criteria for the study

Please note that Physician consent is requisite for the Patient to be enrolled as a participant in the study.

Exclusion Criteria:

1. Major cognitive deficits or psychiatric problems hampering a self-reported evaluation
2. Having received any CML treatment prior to therapy with imatinib, dasatinib, bosutinib or nilotinib for more than three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Cella, PhD, Principal Investigator — Northwestern University; Fabio Efficace, PhD, Principal Investigator — Fondazione GIMEMA
Locations (16):
- United States (2):
  - Augusta University, Hematology and Oncology, Augusta, Georgia
  - Northwestern University, Robert H. Lurie Comprehensive Cancer Center Comprehensive Cancer Center (RHLCCC), Chicago, Illinois
- Italy (14):
  - Policlinico Sant'Orsola Malpighi - UOC Ematologia - Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO - Azienda Ospedaliera G. Brotzu, Cagliari
  - Milano Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - UOC Oncoematologia - Padiglione Marcora, Milan
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - UOC Ematologia, Napoli
  - Azienda Ospedaliera Universitaria Maggiore della Carità di Novara - SCDU Ematologia, Novara
  - AUSL Reggio Emilia - Arcispedale S. Maria Nuova, IRCSS - SC Ematologia, Reggio Emilia
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università degli Studi "Sapienza" - UOC Ematologia, Roma
  - Ospedale Sant'Eugenio, Roma
  - The GIMEMA Foundation (Italian Group for Adult Hematologic Diseases), Rome
  - Azienda Ospedaliero-Universitario Città della Salute e della Scienza di Torino - Ospedale S. Giovanni Battista Molinette - SC Ematologia, Torino
  - Ospedale Mauriziano Umberto I - Torino - SCDU Ematologia, Torino
  - ASUI di Udine - Presidio Ospedaliero "Santa Maria della Misericordia" - Clinica Ematologica, Udine
  - Azienda Ospedaliera Universitario Integrata di Verona, Policlinico G.B. Rossi - UOC Ematologia, Verona
  - USL 6 - Ospedale San Bortolo - Vicenza, Vicenza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Druker BJ, Sawyers CL, Kantarjian H, Resta DJ, Reese SF, Ford JM, Capdeville R, Talpaz M. Activity of a specific inhibitor of the BCR-ABL tyrosine kinase in the blast crisis of chronic myeloid leukemia and acute lymphoblastic leukemia with the Philadelphia chromosome. N Engl J Med. 2001 Apr 5;344(14):1038-42. doi: 10.1056/NEJM200104053441402. PMID 11287973
- [Background] Druker BJ, Talpaz M, Resta DJ, Peng B, Buchdunger E, Ford JM, Lydon NB, Kantarjian H, Capdeville R, Ohno-Jones S, Sawyers CL. Efficacy and safety of a specific inhibitor of the BCR-ABL tyrosine kinase in chronic myeloid leukemia. N Engl J Med. 2001 Apr 5;344(14):1031-7. doi: 10.1056/NEJM200104053441401. PMID 11287972
- [Background] Rosti G, Castagnetti F, Gugliotta G, Baccarani M. Tyrosine kinase inhibitors in chronic myeloid leukaemia: which, when, for whom? Nat Rev Clin Oncol. 2017 Mar;14(3):141-154. doi: 10.1038/nrclinonc.2016.139. Epub 2016 Oct 18. PMID 27752053
- [Background] Cella D, Nowinski CJ, Frankfurt O. The impact of symptom burden on patient quality of life in chronic myeloid leukemia. Oncology. 2014;87(3):133-47. doi: 10.1159/000362816. Epub 2014 Jul 8. PMID 25012261
- [Background] Bower H, Bjorkholm M, Dickman PW, Hoglund M, Lambert PC, Andersson TM. Life Expectancy of Patients With Chronic Myeloid Leukemia Approaches the Life Expectancy of the General Population. J Clin Oncol. 2016 Aug 20;34(24):2851-7. doi: 10.1200/JCO.2015.66.2866. Epub 2016 Jun 20. PMID 27325849
- [Background] Efficace F, Baccarani M, Breccia M, Cottone F, Alimena G, Deliliers GL, Barate C, Specchia G, Di Lorenzo R, Luciano L, Turri D, Martino B, Stagno F, Dabusti M, Bergamaschi M, Leoni P, Simula MP, Levato L, Fava C, Veneri D, Sica S, Rambaldi A, Rosti G, Vignetti M, Mandelli F. Chronic fatigue is the most important factor limiting health-related quality of life of chronic myeloid leukemia patients treated with imatinib. Leukemia. 2013 Jul;27(7):1511-9. doi: 10.1038/leu.2013.51. Epub 2013 Feb 18. PMID 23417029
- [Background] Guerin A, Chen L, Ionescu-Ittu R, Marynchenko M, Nitulescu R, Hiscock R, Keir C, Wu EQ. Impact of low-grade adverse events on health-related quality of life in adult patients receiving imatinib or nilotinib for newly diagnosed Philadelphia chromosome positive chronic myelogenous leukemia in chronic phase. Curr Med Res Opin. 2014 Nov;30(11):2317-28. doi: 10.1185/03007995.2014.944973. Epub 2014 Aug 5. PMID 25025755
- [Background] Williams LA, Garcia Gonzalez AG, Ault P, Mendoza TR, Sailors ML, Williams JL, Huang F, Nazha A, Kantarjian HM, Cleeland CS, Cortes JE. Measuring the symptom burden associated with the treatment of chronic myeloid leukemia. Blood. 2013 Aug 1;122(5):641-7. doi: 10.1182/blood-2013-01-477687. Epub 2013 Jun 18. PMID 23777764
- [Background] Noens L, Hensen M, Kucmin-Bemelmans I, Lofgren C, Gilloteau I, Vrijens B. Measurement of adherence to BCR-ABL inhibitor therapy in chronic myeloid leukemia: current situation and future challenges. Haematologica. 2014 Mar;99(3):437-47. doi: 10.3324/haematol.2012.082511. PMID 24598855
- [Background] Marin D, Bazeos A, Mahon FX, Eliasson L, Milojkovic D, Bua M, Apperley JF, Szydlo R, Desai R, Kozlowski K, Paliompeis C, Latham V, Foroni L, Molimard M, Reid A, Rezvani K, de Lavallade H, Guallar C, Goldman J, Khorashad JS. Adherence is the critical factor for achieving molecular responses in patients with chronic myeloid leukemia who achieve complete cytogenetic responses on imatinib. J Clin Oncol. 2010 May 10;28(14):2381-8. doi: 10.1200/JCO.2009.26.3087. Epub 2010 Apr 12. PMID 20385986
- [Background] Noens L, van Lierde MA, De Bock R, Verhoef G, Zachee P, Berneman Z, Martiat P, Mineur P, Van Eygen K, MacDonald K, De Geest S, Albrecht T, Abraham I. Prevalence, determinants, and outcomes of nonadherence to imatinib therapy in patients with chronic myeloid leukemia: the ADAGIO study. Blood. 2009 May 28;113(22):5401-11. doi: 10.1182/blood-2008-12-196543. Epub 2009 Apr 6. PMID 19349618
- [Background] Ibrahim AR, Eliasson L, Apperley JF, Milojkovic D, Bua M, Szydlo R, Mahon FX, Kozlowski K, Paliompeis C, Foroni L, Khorashad JS, Bazeos A, Molimard M, Reid A, Rezvani K, Gerrard G, Goldman J, Marin D. Poor adherence is the main reason for loss of CCyR and imatinib failure for chronic myeloid leukemia patients on long-term therapy. Blood. 2011 Apr 7;117(14):3733-6. doi: 10.1182/blood-2010-10-309807. Epub 2011 Feb 23. PMID 21346253
- [Background] Efficace F, Cannella L. The value of quality of life assessment in chronic myeloid leukemia patients receiving tyrosine kinase inhibitors. Hematology Am Soc Hematol Educ Program. 2016 Dec 2;2016(1):170-179. doi: 10.1182/asheducation-2016.1.170. PMID 27913477
- [Background] Experts in Chronic Myeloid Leukemia. The price of drugs for chronic myeloid leukemia (CML) is a reflection of the unsustainable prices of cancer drugs: from the perspective of a large group of CML experts. Blood. 2013 May 30;121(22):4439-42. doi: 10.1182/blood-2013-03-490003. Epub 2013 Apr 25. PMID 23620577
- [Background] Kotronoulas G, Kearney N, Maguire R, Harrow A, Di Domenico D, Croy S, MacGillivray S. What is the value of the routine use of patient-reported outcome measures toward improvement of patient outcomes, processes of care, and health service outcomes in cancer care? A systematic review of controlled trials. J Clin Oncol. 2014 May 10;32(14):1480-501. doi: 10.1200/JCO.2013.53.5948. Epub 2014 Apr 7. PMID 24711559
- [Background] Velikova G, Booth L, Smith AB, Brown PM, Lynch P, Brown JM, Selby PJ. Measuring quality of life in routine oncology practice improves communication and patient well-being: a randomized controlled trial. J Clin Oncol. 2004 Feb 15;22(4):714-24. doi: 10.1200/JCO.2004.06.078. PMID 14966096
- [Background] Efficace F, Gaidano G, Lo-Coco F. Patient-reported outcomes in hematology: is it time to focus more on them in clinical trials and hematology practice? Blood. 2017 Aug 17;130(7):859-866. doi: 10.1182/blood-2017-03-737403. Epub 2017 Jul 10. PMID 28694324
- [Background] Efficace F, Baccarani M, Rosti G, Cottone F, Castagnetti F, Breccia M, Alimena G, Iurlo A, Rossi AR, Pardini S, Gherlinzoni F, Salvucci M, Tiribelli M, Vignetti M, Mandelli F. Investigating factors associated with adherence behaviour in patients with chronic myeloid leukemia: an observational patient-centered outcome study. Br J Cancer. 2012 Sep 4;107(6):904-9. doi: 10.1038/bjc.2012.348. Epub 2012 Aug 7. PMID 22871884
- [Background] Dueck AC, Mendoza TR, Mitchell SA, Reeve BB, Castro KM, Rogak LJ, Atkinson TM, Bennett AV, Denicoff AM, O'Mara AM, Li Y, Clauser SB, Bryant DM, Bearden JD 3rd, Gillis TA, Harness JK, Siegel RD, Paul DB, Cleeland CS, Schrag D, Sloan JA, Abernethy AP, Bruner DW, Minasian LM, Basch E; National Cancer Institute PRO-CTCAE Study Group. Validity and Reliability of the US National Cancer Institute's Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). JAMA Oncol. 2015 Nov;1(8):1051-9. doi: 10.1001/jamaoncol.2015.2639. PMID 26270597
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Weidle PJ, Wamai N, Solberg P, Liechty C, Sendagala S, Were W, Mermin J, Buchacz K, Behumbiize P, Ransom RL, Bunnell R. Adherence to antiretroviral therapy in a home-based AIDS care programme in rural Uganda. Lancet. 2006 Nov 4;368(9547):1587-94. doi: 10.1016/S0140-6736(06)69118-6. PMID 17084759
- [Background] Kripalani S, Risser J, Gatti ME, Jacobson TA. Development and evaluation of the Adherence to Refills and Medications Scale (ARMS) among low-literacy patients with chronic disease. Value Health. 2009 Jan-Feb;12(1):118-23. doi: 10.1111/j.1524-4733.2008.00400.x. PMID 19911444
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Phillips KM, Pinilla-Ibarz J, Sotomayor E, Lee MR, Jim HS, Small BJ, Sokol L, Lancet J, Tinsley S, Sweet K, Komrokji R, Jacobsen PB. Quality of life outcomes in patients with chronic myeloid leukemia treated with tyrosine kinase inhibitors: a controlled comparison. Support Care Cancer. 2013 Apr;21(4):1097-103. doi: 10.1007/s00520-012-1630-5. Epub 2012 Nov 20. PMID 23179489
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Basch E, Iasonos A, Barz A, Culkin A, Kris MG, Artz D, Fearn P, Speakman J, Farquhar R, Scher HI, McCabe M, Schrag D. Long-term toxicity monitoring via electronic patient-reported outcomes in patients receiving chemotherapy. J Clin Oncol. 2007 Dec 1;25(34):5374-80. doi: 10.1200/JCO.2007.11.2243. PMID 18048818
- [Background] Baccarani M, Deininger MW, Rosti G, Hochhaus A, Soverini S, Apperley JF, Cervantes F, Clark RE, Cortes JE, Guilhot F, Hjorth-Hansen H, Hughes TP, Kantarjian HM, Kim DW, Larson RA, Lipton JH, Mahon FX, Martinelli G, Mayer J, Muller MC, Niederwieser D, Pane F, Radich JP, Rousselot P, Saglio G, Saussele S, Schiffer C, Silver R, Simonsson B, Steegmann JL, Goldman JM, Hehlmann R. European LeukemiaNet recommendations for the management of chronic myeloid leukemia: 2013. Blood. 2013 Aug 8;122(6):872-84. doi: 10.1182/blood-2013-05-501569. Epub 2013 Jun 26. PMID 23803709
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] O'Brien S, Berman E, Borghaei H, Deangelo DJ, Devetten MP, Devine S, Erba HP, Gotlib J, Jagasia M, Moore JO, Mughal T, Pinilla-Ibarz J, Radich JP, Shah Md NP, Shami PJ, Smith BD, Snyder DS, Tallman MS, Talpaz M, Wetzler M; National Comprehensive Cancer Network. NCCN clinical practice guidelines in oncology: chronic myelogenous leukemia. J Natl Compr Canc Netw. 2009 Oct;7(9):984-1023. doi: 10.6004/jnccn.2009.0065. No abstract available. PMID 19878641
- [Background] Sokal JE, Cox EB, Baccarani M, Tura S, Gomez GA, Robertson JE, Tso CY, Braun TJ, Clarkson BD, Cervantes F, et al. Prognostic discrimination in "good-risk" chronic granulocytic leukemia. Blood. 1984 Apr;63(4):789-99. PMID 6584184
- [Background] Alonso J, Bartlett SJ, Rose M, Aaronson NK, Chaplin JE, Efficace F, Leplege A, Lu A, Tulsky DS, Raat H, Ravens-Sieberer U, Revicki D, Terwee CB, Valderas JM, Cella D, Forrest CB; PROMIS International Group. The case for an international patient-reported outcomes measurement information system (PROMIS(R)) initiative. Health Qual Life Outcomes. 2013 Dec 20;11:210. doi: 10.1186/1477-7525-11-210. PMID 24359143
- [Background] Cottone F, Deliu N, Collins GS, Anota A, Bonnetain F, Van Steen K, Cella D, Efficace F. Modeling strategies to improve parameter estimates in prognostic factors analyses with patient-reported outcomes in oncology. Qual Life Res. 2019 May;28(5):1315-1325. doi: 10.1007/s11136-018-02097-2. Epub 2019 Jan 18. PMID 30659449
- [Background] Efficace F, Baccarani M, Breccia M, Saussele S, Abel G, Caocci G, Guilhot F, Cocks K, Naeem A, Sprangers M, Oerlemans S, Chie W, Castagnetti F, Bombaci F, Sharf G, Cardoni A, Noens L, Pallua S, Salvucci M, Nicolatou-Galitis O, Rosti G, Mandelli F. International development of an EORTC questionnaire for assessing health-related quality of life in chronic myeloid leukemia patients: the EORTC QLQ-CML24. Qual Life Res. 2014 Apr;23(3):825-36. doi: 10.1007/s11136-013-0523-5. Epub 2013 Sep 13. PMID 24026634
- [Derived] Efficace F, Cottone F, Yanez B, Kota V, Castagnetti F, Caocci G, Bonifacio M, Patriarca A, Capodanno I, Miggiano MC, Tiribelli M, Breccia M, Luciano L, Giai V, Iurlo A, Abruzzese E, Fava C, Dinner S, Altman JK, Rosti G, Cortes J, Vignetti M, Cella D. Patient-reported symptom monitoring and adherence to therapy in patients with newly diagnosed chronic myeloid leukemia. Cancer. 2024 Jan;130(2):287-299. doi: 10.1002/cncr.35021. Epub 2023 Oct 6. PMID 37801052
- See also: FACIT Searchable Library and Custom Form Developer (Build-a-PRO) — https://wizard.facit.org
- See also: EORTC Quality of Life Group Item Library — https://www.eortc.be/itemlibrary/

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Myeloid Leukemia (CML) Patients: CML patients undergoing first-line tyrosine kinase inhibitor (TKI) therapy
  EMPATHY Pilot: The goal of this pilot is to develop and pilot a tailored monitoring intervention targeting symptomatic, Patient-reported adverse events (AEs) in chronic myeloid leukemia (CML) Patients undergoing first-line tyrosine kinase inhibitor (TKI) therapy. The tailored monitoring intervention will draw primarily from the Patient Reported Outcome (PRO-CTCAE) Item Library, with additional items drawn from the FACIT and EORTC Item libraries as necessary. After identifying the full set of AEs to be monitored, we will load the Patient assessment and report program into tablets for electronic administration in the busy clinic setting. We will then pilot a six-month intervention aimed to monitor and manage emerging AEs, coupled with assessment of intervention feasibility, Patient acceptability and satisfaction, provider acceptability and clinical management utility, adherence to TKI therapy, and HRQoL. We expect that adherence to therapy, clinical response, and HRQoL will be enhanced by such an intervention.
Period: Overall Study
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Started | 94
Completed | 90
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Although 94 participants were consented, one participant withdrew before baseline, so we have 93 participants with data
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.92 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 81
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 16
  Italy | 78

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: Adherence to Refills and Medications Scale (ARMS). The ARMS-7 consists of seven items evaluating adherence to taking medications and refilling prescriptions. Items are rated on a four-point Likert scale ranging between 7 and 28, with higher scores indicating lower medication adherence.
Time Frame: 6 months
Population: 94 patients were consented. 93 patients provided baseline information. 83 patients provided adherence outcome data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Number analyzed (Participants) | 83
score on a scale | 7.81 (1.31)

2. Primary Outcome: Number of Participants Adherent To Their Medication
Description: Prescription refill data extracted from hospital pharmacy records. Prescription refill data were evaluated over 6 months. Missed refills, for reasons other than mortality or physician change of medication, were counted as non-adherence. Adherence was defined as the number of days medicine not available between each refill over the number of days between first prescription and last refill during the study period.
Time Frame: 6 months
Population: although 94 patients signed consent, one withdrew prior to baseline and so the number of participants analyzed is 93
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Number analyzed (Participants) | 93
Participants | 86

3. Secondary Outcome: Health-Related Quality of Life
Description: Functional Assessment of Cancer Therapy-General. The possible score range of this measure is 0-128. Higher scores denote better quality of life
Time Frame: 6 months
Population: 94 patients were consented. 93 patients provided baseline information. 84 patients provided adherence outcome data
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Number analyzed (Participants) | 84
score on a scale | 81.4 [78.4 to 84.3]

4. Secondary Outcome: Fatigue
Description: Functional Assessment of Chronic Illness Therapy-Fatigue. the possible score range of this measure is 0-52. Higher scores reflect less fatigue
Time Frame: 6 months
Population: 94 patients were consented. 93 patients provided baseline information. 84 patients provided adherence outcome data
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Number analyzed (Participants) | 84
score on a scale | 41.9 [40 to 43.8]

5. Secondary Outcome: Cytogenetic Response
Description: Cytogenetic response (CyR) is defined based on the percentage of Ph pos metaphases, as evaluated by chromosome banding analysis of at least 20 marrow cell metaphases (cytogenetics). Complete CyR is when the percentage of Ph pos metaphases is 0; Partial CyR is when the percentage of Ph pos metaphases ranges from 1 to 35, Minor CyR if the percentage of Ph pos metaphases ranges from 36 to 65, minimal CyR if the percentage of Ph pos metaphases ranges from 66 to 95, No CyR if the percentage of Ph pos metaphases is higher than 95.
Time Frame: 6 months
Population: 94 patients were consented. 93 patients provided baseline information. 81 patients provided adherence outcome data
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
Number analyzed (Participants) | 81
Participants | 61

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Chronic Myeloid Leukemia (CML) Patients
All-Cause Mortality (participants affected / at risk) | 1/94
Serious Adverse Events (participants affected / at risk) | 13/94
Other Adverse Events (participants affected / at risk) | 0/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Myeloid Leukemia (CML) Patients (N=94)
abdominal pain (Gastrointestinal disorders) | 1
Neutropenia (Immune system disorders) | 5
thrombocytopenia (Blood and lymphatic system disorders) | 4
neutropenia (Immune system disorders) | 6
myocardial infarction (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT04384848/Prot_SAP_000.pdf